CLINICAL TRIAL: NCT06237621
Title: Study to Use Change in Near Infrared Spectroscopy Assessment of Tissue Oxygenation During a Provocative Leg Maneuver to Assess Peripheral Artery Disease State.
Brief Title: Using SnapshotNIR With Provocative Leg Maneuver for PAD Assessment
Status: Recruiting | Type: Observational
Sponsor: Kent Imaging Inc (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 20230638HU
Record Dates: First submitted 2024-01-10; First posted 2024-02-01 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Ankle-brachial index; Tissue Oxygen Saturation; Near infrared spectroscopy; NIR; Peripheral Arterial Disease; PAD; CLI; Provocative Leg Maneuver; PAD screening
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- People at risk of PAD
  Interventions: Device: SnapshotNIR imaging

INTERVENTIONS:
Device: SnapshotNIR imaging — SnapshotNIR will be used for tissue oxygen-saturation imaging of all the subjects' foot along with standard of care procedures for PAD assessment.

SUMMARY:
The objective of this trial is to determine if Near-infrared spectroscopy (NIRS) can accurately evaluate the degree of Peripheral Arterial Disease (PAD) during a Provocative Elevation Maneuver of the Lower Extremity (PEMLE) test, as compared to routine clinical assessments.

DETAILED DESCRIPTION:
This study is designed as a prospective observational study to assess the effectiveness of NIRS to accurately evaluate the degree of PAD, as compared to routine clinical assessment, during the PEMLE test protocol. This will be a single visit study where subjects will be screened and enrolled during a regular clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* 35-99 years of age
* Subject has at least 1 intact forefoot
* Can achieve leg positions to complete the study

Exclusion Criteria:

* The subject is unwilling or unable to comply with the protocol or scheduled appointments.
* The subject has had transmetatarsal amputation or higher on both limbs.
* Vascular intervention within the past year
* Subjects who have had a previous distal bypass procedure
* Pregnant or plans to become pregnant
* Deemed by the PI to be unsuitable for the study

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled through the PI's clinic population. Healthy volunteers will be recruited from the clinic staff population and other volunteers recruited from healthy clinic visitors. Subjects who are identified for study participation will be screened for all eligibility requirements. Those meeting eligibility criteria for the study will have the study explained to them by the study staff. An Informed Consent Form will be provided to sign, prior to undergoing any study procedures. Subjects will be encouraged to ask questions of the study staff. There is no cap on the number of subjects that can be screened. Additional subjects will continue to be recruited as needed to reach the total study enrollment of 250 limbs.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparing change in plantar foot NIRS measurements (baseline vs raised position) during a Provocative Maneuver Leg Raise test to the SOC clinical assessment of PAD | 1-2 days
  The significance of the relationship will be evaluated using an analysis of variance (ANOVA) where the independent variable will be the SOC assessment of PAD and the dependent variable will be the difference in NIRS measurement between the initial position (supine) and the second position (elevated leg).

SECONDARY OUTCOMES:
Comparing change in plantar foot NIRS measurements (baseline vs raised position) during a Provocative Maneuver Leg Raise test paired with the presence/absence of diabetes to the SOC clinical assessment of PAD | 1-2 days
  This outcome will be evaluated using an analysis of variance (ANOVA) with two independent variables (factors) including the SOC assessment of PAD and the presence of diabetes (present or not) and the dependent variable will be the difference in NIRS measurement between the initial position (supine) and the second position (elevated leg).
Comparing change in dorsal foot NIRS measurements (baseline vs raised position) during a Provocative Maneuver Leg Raise test to the SOC clinical assessment of PAD | 1-2 days
  This outcome will be evaluated in a similar fashion as the analysis from the primary outcome but with the dependent variable will be calculated based on measurements taken from the dorsal surface of the foot which will be evaluated against the independent variable (SOC assessment) via ANOVA.
Change of NIRS measurements with other positions | 1-2 days
  This outcome will be evaluated in a similar fashion as the analysis from the primary outcome but with the dependent variable being the difference in NIRS measurement between the raised and dependent position (patient sitting up) and then the baseline and dependent position which will be evaluated against the independent variable (SOC assessment) via ANOVA.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No